CLINICAL TRIAL: NCT04702763
Title: Eye Movements Recording Using a Smartphone: Comparison to Standard Video-oculography Data in Patients With Multiple Sclerosis
Brief Title: Eye Movements Recording Using a Smartphone: Comparison to Standard Video-oculography in Patients With Multiple Sclerosis
Status: Completed | Type: Observational
Sponsor: Association de Recherche Bibliographique pour les Neurosciences (Other)
Collaborators: Centre Hospitalier Princesse Grace (Other); Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: e-VOG
Record Dates: First submitted 2021-01-07; First posted 2021-01-11 (Actual); Last update posted 2022-01-27 (Actual); Status verified 2022-01

CONDITIONS: Multiple Sclerosis
Keywords: Demyelinating disease; Multiple Sclerosis; Video-oculography; Eye-Tracking; Eye movements; Subclinical oculomotor abnormalities; Oculomotor disorders
MeSH Terms: conditions — Multiple Sclerosis; Demyelinating Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Multiple Sclerosis (Eye-Tracker®T2 + e-VOG): Multiple Sclerosis subjects who first perform standard video-oculography assessment, followed by e-VOG digital assessment.
  Interventions: Other: Eye-Tracker®T2 + e-VOG
- Multiple Sclerosis (e-VOG + Eye-Tracker®T2): Multiple Sclerosis subjects who first perform e-VOG digital assessment, followed by the standard video-oculography assessment.
  Interventions: Other: e-VOG + Eye-Tracker®T2

INTERVENTIONS:
Other: Eye-Tracker®T2 + e-VOG — * 1st step: eyes movements assessed with standard video-oculography device
  * 2° step: eyes movements assessed with e-VOG digital application
  * Patient study duration is about 30 minutes, the day the patient performs their standard video-oculography examination in routine care
  Groups: Multiple Sclerosis (Eye-Tracker®T2 + e-VOG)
Other: e-VOG + Eye-Tracker®T2 — * 1st step: eyes movements assessed with e-VOG digital application
  * 2° step: eyes movements assessed with standard video-oculography device
  * Patient study duration is about 30 minutes, the day the patient performs their standard video-oculography examination in routine care
  Groups: Multiple Sclerosis (e-VOG + Eye-Tracker®T2)

SUMMARY:
This study aims to compare measurements obtained through the e-VOG application (mobile application, usable on mobile phones or tablets, to measure eye movements) with measurements from the standard video-oculography device (Eye-Tracker®T2), in patient with Multiple Sclerosis.

DETAILED DESCRIPTION:
Based on literature, investigators hypothesize that it would be relevant to focus more broadly on subclinical abnormalities of oculomotricity in multiple sclerosis (MS). However, the difficulty of accessing video-oculography platforms (or eye-tracking devices) is probably one of the main limitations to performing this type of assessment.

To respond this problem, the "Resources and Skills Center-Multiple Sclerosis" (CRC SEP) team at the Nice University Hospital Center (France) has developed a mobile application (named e-VOG), usable on mobile phones or tablets, to measure eye movements. e-VOG reproduces the classic paradigms of video-oculography to collect data similar to standard video-oculography recording (saccade latency and speed, anti-saccade error rate, presence of fixation abnormalities).

e-VOG will not replace standard video-oculography platforms, because its technical characteristics are not as high. But investigators hypothesize that this application could constitute a screening tool for subclinical oculomotor abnormalities, usable by neurologists in consultation, directly on their mobile, which would make it possible to select a smaller population of patients in whom a further exploration by standard video-oculography would be indicated.

Memory Center of the Rainier III Gerontologic Center (Princess Grace Hospital - Monaco) is equipped with a standard video-oculography device, also named eye-tracking device (Eye-Tracker®T2), which records eye movements at a high frequency and measures saccades parameters (latency, speed, amplitudes etc...).

This study is a collaborative study between the Center Rainier III team and the CRC SEP team in Nice. Its objective will be to compare measurements obtained through the e-VOG application with measurements from the standard video-oculography device.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female.
* 18 years old and above.
* referred by a neurologist to perform a video-oculography (Eye-Tracking) examination as part of routine care.
* with Multiple Sclerosis (defined according to McDonald's 2017 criteria).
* covered by a health insurance system
* volunteer, able to give free, informed and written consent.

Exclusion Criteria:

* General anaesthesia within 3 months.
* Neurological, ophthalmological or general pathology preventing the realization of a video-oculography examination.
* Oculomotor abnormality detectable on clinical examination by the neurologist prescribing the standard video-oculography examination.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from patients with MS for whom a standard video-oculography exam is prescribed by the CRC SEP of the CHU de Nice (France) as part of routine care.
  Standard video-oculography exam is carried out at the Center Rainier III (Princess Grace Hospital - Monaco), in accordance with usual practices. It is used at the Centre Rainier III since August 2014. It is a non-invasive device for eye movements recording, allowing doctors and researchers to measure standard parameters related to eye movements. Developed by the Eye Brain Company (France), this is a Class IIa medical device, CE marking, according to Annexe IX of the directive 93/42/CE
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2020-10-08 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2021-10-30 (Actual)

PRIMARY OUTCOMES:
Oculomotor profiles concordance | Day 0
  Analyze of the concordance of the profiles obtained between the e-VOG digital assessment and the standard video-oculography assessment.
  Evaluation criteria: For each assessment, patients will be classified into 3 profiles (Profile 1 = profile without oculomotor abnormality; Profile 2 = intermediate profile with 1 to 2 oculomotor abnormalities; Profile 3: profile with 3 to 4 oculomotor anomalies), based on the observation of 4 parameters (latency / speed / fixation disorders / presence of internuclear ophthalmoplegia), in accordance with the literature standards.

SECONDARY OUTCOMES:
Latency during horizontal reflex saccades | Day 0
  Measure of Latency during an horizontal reflex saccades paradigm with e-VOG Compared to the one performed with standard video-oculography device.
  Evaluation criteria: latency (reaction time in ms).
Latency during vertical reflex saccades | Day 0
  Measure of Latency during a vertical reflex saccades paradigm with e-VOG Compared to the one performed with standard video-oculography device.
  Evaluation criteria: latency (reaction time in ms).
Velocity during horizontal reflex saccades | Day 0
  Measure of Velocity during an horizontal reflex saccades paradigm with e-VOG Compared to the one performed with standard video-oculography device.
  Evaluation criteria: velocity (mean and peak velocity) in °/s.
Velocity during vertical reflex saccades | Day 0
  Measure of Velocity during a vertical reflex saccades paradigm with e-VOG Compared to the one performed with standard video-oculography device.
  Evaluation criteria: velocity (mean and peak velocity) in °/s.
Inhibition capacity | Day 0
  Measure of inhibition capacity performance during an antisaccades" paradigm with e-VOG Compared to the one evaluated with standard video-oculography device.
  Evaluation criteria: percentage of errors.
Internuclear ophthalmoplegia (INO) detection | Day 0
  Highlight presence/absence of INO with e-VOG Compared to standard video-oculography device.
  Evaluation criteria: INO is present if calculated ratio of abducting to adducting eye movement (both mean and peak velocity) is >1.
Fixations impairments detection | Day 0
  Highlight presence/absence of Fixations impairments with e-VOG Compared to standard video-oculography device.
  Evaluation criteria: presence/absence/frequency of square wave-jerks, nystagmus, flutters.
Impairment of horizontal smooth pursuit | Day 0
  Highlight Impairment of horizontal smooth pursuit with e-VOG Compared to standard video-oculography device.
  Evaluation criteria: presence/absence of saccade and perturbation.
Impairment of vertical smooth pursuit | Day 0
  Highlight Impairment of horizontal smooth pursuit with e-VOG Compared to standard video-oculography device.
  Evaluation criteria: presence/absence of saccade and perturbation.
Patient acceptability of the e-VOG digital assessment | Day 0
  Comparison of patient acceptability between the e-VOG digital assessment and the standard video-oculography assessment.
  Evaluation criteria: satisfaction questionnaire given to the patient at the end of assessments. 2 questions on the difficulty or discomfort felt during the 2 assessments.

CONTACTS AND LOCATIONS:
Overall Officials: Mikael COHEN, MD, Principal Investigator — Centre de Ressources et de Compétences SEP, UMRC Pasteur 2, Université Nice Côte d'Azur, Nice-France; Christine LEBRUN-FRENAY, PUPH, Principal Investigator — Centre de Ressources et de Compétences SEP, UMRC Pasteur 2, Université Nice Côte d'Azur, Nice-France; Sandrine LOUCHART DE LA CHAPELLE, MD-PHD, Principal Investigator — Centre Mémoire, Centre de Gérontologie Clinique RAINIER III, Princess Grace Hospital, Monaco; Alain PESCE, PUPH, Study Director — AREBISN (Association de Recherche Bibliographique pour les Neurosciences), Nice (France)
Locations (1):
- Centre Mémoire / Centre de Gérontologie Clinique Rainier III / Princess Grace Hospital, Monaco, Monaco

IPD SHARING:
Plan to Share IPD: No